CLINICAL TRIAL: NCT00163488
Title: Investigation of Potential Additive Inhibitory Effects on HPA-Axis of Ciclesonide Nasal Spray When Administered Concomitantly With Orally Inhaled Fluticasone Propionate/Salmeterol (FP/SAL) in Patients (18-60 Years) With Perennial Allergic Rhinitis (PAR)
Brief Title: Safety of Ciclesonide Nasal Spray Administered With Inhaled Fluticasone Dipropionate/Salmeterol in Adults With Perennial Allergic Rhinitis (BY9010/M1-409)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-409
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Perennial Allergic Rhinitis; Allergic Rhinitis; Hay Fever
Keywords: Allergy; Perennial Allergic Rhinitis; Allergic Rhinitis; Hay Fever
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic; Rhinitis, Allergic, Seasonal; Hypersensitivity | interventions — ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of combined ciclesonide nasal spray administered along with a fixed combination of inhaled fluticasone dipropionate/salmeterol.

ELIGIBILITY:
Main Inclusion Criteria:

* General good health, other than perennial allergic rhinitis
* History and diagnosis of perennial allergic rhinitis by skin prick
* Normal body weight as defined by the study protocol

Main Exclusion Criteria:

* Pregnancy, nursing, or plans to become pregnant or donate gametes (ova or sperm) for in vitro fertilization during the study period or for 30 days following the study period
* Participation in any investigational drug trial within the 30 days preceding the Screening Visit
* A known hypersensitivity to any corticosteroid or any of the excipients in the formulations
* Use of any prohibited concomitant medications as defined by the study protocol
* Previous participation in an intranasal ciclesonide study
* Non-vaccinated exposure to or active infection with, chickenpox or measles within the 21 days preceding the Screening Visit

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106
Dates: Start 2005-01; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
safety.

SECONDARY OUTCOMES:
safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Altana Pharma/Nycomed, Long Beach, California, United States

REFERENCES:
- See also: BY9010-M1-409-RDS-2005-12-12.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4537&filename=BY9010-M1-409-RDS-2005-12-12.pdf